CLINICAL TRIAL: NCT01324271
Title: A Clinical Study Of The Acclarent Tympanostomy Tube (Tula™) Delivery System In-Office
Brief Title: inVENT-In-Office Study
Acronym: inVENT-IO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR005016
Record Dates: First submitted 2011-03-23; First posted 2011-03-29 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media
Keywords: Tympanostomy tube placement
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tympanostomy tube placement (Experimental): placement of tympanostomy tube under local anesthesia in office/clinic setting
  Interventions: Device: Acclarent Tympanostomy Tube Delivery system (TTDS)

INTERVENTIONS:
Device: Acclarent Tympanostomy Tube Delivery system (TTDS) — placement of tympanostomy tube under local anesthesia
  Other Names: Tula™

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of the Acclarent Tympanostomy Tube Delivery System (TTDS) for the placement of tympanostomy tubes (TT) under local anesthesia in an office/clinic setting.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo tympanostomy tube insertion
* At least 6 months old
* Behavioral capacity and cooperative temperament to undergo an awake procedure (based on physician judgement)

Exclusion Criteria:

* History of sensitivity or reaction to anesthesia chosen for the procedure
* Significantly atrophic, bimeric, or completely atelectatic tympanic membrane
* Otitis externa
* Anatomy that precludes sufficient visualization of and access to the tympanic membrane
* Anatomy that necessitates tympanostomy tube placement in the posterior half of the tympanic membrane

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Lead-ins & study cohort included (n=85). Same criteria/procedure for all 85 subjects. Study phases did not have different start/end dates. Periods/dates for lead-ins & cohort not different. Physicians with no TTDS experience were required to perform lead-ins in OR (n=26/85). Sites on-boarded and completed lead-ins at different times.
Groups:
- Tympanostomy Tube Placement (Lead-In Procedures): Acclarent Tympanostomy Tube Delivery system (TTDS):
  Placement of tympanostomy tube under local anesthesia in office/clinic setting or under general anesthesia in operating room.
- Tympanostomy Tube Placement (Study Cohort): Acclarent Tympanostomy Tube Delivery system (TTDS): Placement of tympanostomy tube under local anesthesia in office/clinic setting
Period: Overall Study
Arm/Group | Tympanostomy Tube Placement (Lead-In Procedures) | Tympanostomy Tube Placement (Study Cohort)
Started | 57 | 28
Completed | 53 | 28
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Fifty-nine (59) subjects were treated with TTDS in the office under local anesthesia, and 26 were treated with TTDS in the OR under general anesthesia.
Groups:
- Tympanostomy Tube Placement: All enrolled subjects for which a tympanostomy tube was attempted to be placed using a Tympanostomy Tube Delivery System (TTDS) under local anesthesia in office/clinical setting.
Arm/Group | Tympanostomy Tube Placement
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.01 (24.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 45
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 9
  White | 62
  Asian | 1
  Other races (self-reported) | 13
Region of Enrollment [Number; unit: participants]
  United States | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With In-office Tube Placement Procedure Success
Description: Procedure Success is defined as the successful placement of any tympanostomy tube in all enrolled ears in a given subject. Procedure Success is determined on a per subject basis: the rate was calculated based on the number of subjects achieving Procedure Success out of the total number of enrolled subjects. Only subjects for whom tubes were placed under local anesthesia were evaluated for Procedure Success.
Time Frame: Day 0
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Tympanostomy Tube Placement
Number analyzed (Participants) | 59
Percentage of Subjects | 93.2 [83.5 to 98.1]

2. Primary Outcome: Percentage of Tubes Successfully Placed Using a TTDS Device
Description: Device (TTDS) success is defined as the successful delivery of a pre-loaded TT tube across the tympanic membrane using the TTDS. Device success will be evaluated per device attempted. Office/clinical subjects only.
  A Device (Type of Unit analyzed) is defined as a TDS attempt. This is not synonymous with "tube." Tube is the outcome of the device use.
Time Frame: Day 0
Population: All enrolled subjects for which a tympanostomy tube was attempted to be placed using a Tympanostomy Tube Delivery System (TTDS) under local anesthesia in office/clinical setting
Measure: Number (95% Confidence Interval); unit: percentage of devices
Units Other Than Participants: TTDS devices
Groups:
- Tube Placement Using the TTDS in Office/Clinic Setting: All enrolled subjects for which a tympanostomy tube was attempted to be placed using a Tympanostomy Tube Delivery System (TTDS) under local anesthesia in office/clinical setting
Arm/Group | Tube Placement Using the TTDS in Office/Clinic Setting
Number analyzed (Participants) | 59
Number analyzed (TTDS devices) | 90
percentage of devices | 82.2 [72.7 to 89.5]

3. Secondary Outcome: Number of Retained (TTDS-placed) Tubes
Description: Tube retention is the presence of a TT placed successfully by the TTDS device across the tympanic membrane at the two week follow-up visit. Tube retention was confirmed by physician investigator evaluation. N=74 tubes were successfully placed intraprocedurally. Analysis population includes office/clinical subjects only.
Time Frame: 14 days
Population: Total in-office (IO) subjects.
Measure: Number; unit: tubes
Units Other Than Participants: tubes placed via TTDS
Arm/Group | Tympanostomy Tube Placement
Number analyzed (Participants) | 59
Number analyzed (tubes placed via TTDS) | 74
tubes | 74

ADVERSE EVENTS:
Time Frame: 2 weeks post-procedure
Groups:
- Tympanostomy Tube Placement: All enrolled subjects for which a tympanostomy tube was attempted to be placed using a Tympanostomy Tube Delivery System (TTDS).
Arm/Group | Tympanostomy Tube Placement
Serious Adverse Events (participants affected / at risk) | 1/85
Other Adverse Events (participants affected / at risk) | 18/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tympanostomy Tube Placement (N=85)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) — Not device or procedure related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tympanostomy Tube Placement (N=85)
Occluded TT (Ear and labyrinth disorders) | 7 (7)
Otalgia (Ear and labyrinth disorders) | 3 (3)
Otitis Media (Ear and labyrinth disorders) | 2 (2)
Otorrhea (Ear and labyrinth disorders) | 1 (1)
Aural Fullness (Ear and labyrinth disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — not device or procedure related
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — not device or procedure related
Gastroenteritis (Gastrointestinal disorders) | 1 (1) — not device or procedure related
Tube Medialization (Ear and labyrinth disorders) | 1 (1) — re-positioned during procedure with no sequelae

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days